CLINICAL TRIAL: NCT06346028
Title: A Pragmatic Feasibility Trial on the Implementation of Transcranial Magnetic Stimulation for Smoking Cessation
Brief Title: Implementation of Transcranial Magnetic Stimulation for Smoking Cessation
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023/086
Record Dates: First submitted 2024-03-20; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Smoking
Keywords: smoking cessation; quitting smoking; repetitive transcranial magnetic stimulation; rTMS; nicotine dependence
MeSH Terms: conditions — Smoking; Smoking Cessation; Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients Receiving rTMS (Experimental): Participants will receive 3 weeks of daily (Monday to Friday) rTMS sessions followed by 3 weeks of weekly rTMS sessions for a total of 6 weeks of treatment. Each session lasts about 25 minutes and is provided by an rTMS technician at the Temerty Center at 1025 Queen Street West, with medical supervision.
  Interventions: Device: Brainsway H4 deep rTMS coil and Brainsway stimulator system

INTERVENTIONS:
Device: Brainsway H4 deep rTMS coil and Brainsway stimulator system — An rTMS treatment course consisting of daily treatment, 5 days per week, for 3 weeks, followed by once weekly treatments for 3 weeks, for a total of 18 treatment sessions over 6 weeks.
  Sixty trains of 30 pulses each (total 1,800 pulses) will be applied at 10 Hz, for 3 second trains, with a 15 second inter-train interval, for approximately 18 minutes of treatment time.
  At each rTMS treatment session, prior to stimulation, participants will undergo a smoking craving provocation procedure where they will be asked to close their eyes and imagine one of their triggers for 30 seconds. Following this they will watch a PowerPoint presentation of smoking pictures for 2 minutes and 30 seconds. Thus, the entire craving provocation procedure will be 3 minutes prior to stimulation start.
  Brief behavioural support will be available to the participant on a weekly basis by a trained research staff member from the NDC.
  Other Names: Deep rTMS

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) is an alternative non-invasive treatment to help people quit smoking. rTMS uses a magnetic field to stimulate regions of the brain that are involved in addiction. The two brain regions that are stimulated are the insula and the dorsolateral prefrontal cortex, which are involved in drug craving and decision-making, respectively.

The goal of this clinical trial is to learn more about the feasibility of offering rTMS as a treatment in the Nicotine Dependence Clinic (NDC) to help daily smokers to quit smoking. The NDC is at the Center for Addiction and Mental Health (CAMH) at 1025 Queen Street West, in Toronto, Canada.

Participants will be asked to come to CAMH to:

* Complete surveys and optional interviews to learn more about their opinions and experiences with this treatment
* Start a treatment course that includes 3 weeks of daily (Monday to Friday) rTMS sessions followed by 3 weeks of weekly rTMS sessions for a total of 6 weeks. Each session lasts about 25 minutes and is provided by an rTMS technician with medical supervision.

Objectives

• Learning about the feasibility of rTMS as a treatment option for patients in the NDC will help us improve the treatment when offering it in other clinics, which may help improve smoking quit rates and people's overall health.

DETAILED DESCRIPTION:
Approximately 45,000 Canadians die from smoking each year and smoking is the leading preventable cause of death worldwide. Quitting smoking is difficult, and current treatments such as varenicline and nicotine replacement therapy are not always able to help people quit.

Repetitive transcranial magnetic stimulation (rTMS) is an alternative non-invasive treatment to help people quit smoking. rTMS uses a magnetic field to stimulate regions of the brain that are involved in addiction. The two brain regions that are stimulated are the insula and the dorsolateral prefrontal cortex, which are involved in drug craving and decision-making, respectively.

A landmark 2021 study showed that daily rTMS treatment for 6 weeks targeting these regions is effective at reducing craving and cigarette use. This study's findings provided supporting evidence that led Health Canada and the Food and Drug Administration to approve rTMS as a treatment for smoking cessation. Currently, this treatment is not widely available, therefore it is important to learn more about how to bring it into clinics and develop it further.

The goal of this clinical trial is to learn more about the feasibility of offering rTMS as a treatment in the Nicotine Dependence Clinic (NDC) to help daily smokers to quit smoking. The NDC is at the Center for Addiction and Mental Health (CAMH) at 1025 Queen Street West, in Toronto, Canada.

The main questions it aims to answer are:

* How many people who are patients at the NDC are interested in this treatment?
* How acceptable is this treatment for people who have experienced it?
* What factors of this treatment are appealing or unappealing to people?
* How well does it work to help people quit smoking?
* Who are the main group of people who want this treatment?

Participants will be asked to come to CAMH to:

* Complete surveys and optional interviews to learn more about their opinions and experiences with this treatment
* Start a treatment course that includes 3 weeks of daily (Monday to Friday) rTMS sessions followed by 3 weeks of weekly rTMS sessions for a total of 6 weeks. Each session lasts about 25 minutes and is provided by an rTMS technician with medical supervision.

Objectives

• Learning about the feasibility of rTMS as a treatment option for patients in the NDC will help us improve the treatment when offering it in other clinics, which may help improve smoking quit rates and people's overall health.

ELIGIBILITY:
Inclusion Criteria: Patients receiving rTMS

* Smoking cigarettes daily (self-reported)

Inclusion Criteria: Health care providers

* Currently employed as a HCP (physician, social worker, occupational therapist, etc.) at the CAMH NDC
* Involved in the care of at least 1 patient who has received rTMS for smoking cessation

Exclusion Criteria: Patients receiving rTMS

* Have any intracranial implant (e.g., aneurysm clips) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed.
* Pregnant or intending to be pregnant during the study.
* A history of a primary seizure disorder, seizure associated with an intracranial lesion, recurrent seizures related to substance intoxication or withdrawal or recent seizure within the last 6 months.
* Taking any anticonvulsant medication unless it cannot be tapered or discontinued due to risk of clinical safety or destabilization, according to the participant or their referring physician.
* Taking benzodiazepines with dose equivalent or greater than lorazepam 2mg/day unless it cannot be tapered or discontinued due to risk of clinical safety or destabilization, according to the participant or their referring physician.
* Space occupying intracranial lesion.
* Acutely unstable medical, psychiatric, or substance use disorder comorbidity with safety concerns at the discretion of the PI or study physician.

Exclusion Criteria: Health care providers

- There are no exclusion criteria for HCP Participants

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The primary objective of the study is to evaluate the feasibility of implementing rTMS in the Nicotine Dependence Clinic (NDC) at CAMH, in Toronto. This is determine by reach, the extent to which patients are engaging in the rTMS treatment. | Through study completion, an average of 1 year
  The proportion of patients accepting rTMS relative to all patients with a visit to the NDC during the study period.
Identify rates of adoption of rTMS in Nicotine Dependence Clinic | Through study completion, an average of 1 year
  What percentage of NDC HCPs refer patients to rTMS treatment? (Adoption)
Identify contextual determinants of rTMS adoption and reach NDC through a qualitative approach. | Through study completion, an average of 1 year
  Research questions assessed through through surveys and semi-structured interviews
  1. What are the multi-level barriers and facilitators to integrating rTMS in NDC?
  2. How acceptable, appropriate and feasible is it to integrate rTMS in NDC?

SECONDARY OUTCOMES:
Evaluate the effectiveness of rTMS on smoking cessation rates in real world patients with common comorbidities seeking treatment at NDC. | Through study completion, an average of 1 year
  Self-reported 4-week continuous quit rate and long follow-up continuous quit rate (biochemically verified by urine nicotine/tobacco metabolite collection and analysis at end of treatment and the long follow-up).
Explore patient-HCP communication about shared treatment decision-making for rTMS. | Through study completion, an average of 1 year
  We will conduct semi-structured interviews with NDC patients and HCPs to better understand the collaborative nature and necessary communication components involved in shared treatment decision-making for rTMS.

CONTACTS AND LOCATIONS:
Overall Officials: Victor Tang, MD, MSc, Principal Investigator — Center for Addiction and Mental Health
Locations (1):
- Center for Addiction and Mental Health (CAMH), Toronto, Ontario, Canada

REFERENCES:
- [Background] Zangen A, Moshe H, Martinez D, Barnea-Ygael N, Vapnik T, Bystritsky A, Duffy W, Toder D, Casuto L, Grosz ML, Nunes EV, Ward H, Tendler A, Feifel D, Morales O, Roth Y, Iosifescu DV, Winston J, Wirecki T, Stein A, Deutsch F, Li X, George MS. Repetitive transcranial magnetic stimulation for smoking cessation: a pivotal multicenter double-blind randomized controlled trial. World Psychiatry. 2021 Oct;20(3):397-404. doi: 10.1002/wps.20905. PMID 34505368
- [Background] Ekhtiari H, Tavakoli H, Addolorato G, Baeken C, Bonci A, Campanella S, Castelo-Branco L, Challet-Bouju G, Clark VP, Claus E, Dannon PN, Del Felice A, den Uyl T, Diana M, di Giannantonio M, Fedota JR, Fitzgerald P, Gallimberti L, Grall-Bronnec M, Herremans SC, Herrmann MJ, Jamil A, Khedr E, Kouimtsidis C, Kozak K, Krupitsky E, Lamm C, Lechner WV, Madeo G, Malmir N, Martinotti G, McDonald WM, Montemitro C, Nakamura-Palacios EM, Nasehi M, Noel X, Nosratabadi M, Paulus M, Pettorruso M, Pradhan B, Praharaj SK, Rafferty H, Sahlem G, Salmeron BJ, Sauvaget A, Schluter RS, Sergiou C, Shahbabaie A, Sheffer C, Spagnolo PA, Steele VR, Yuan TF, van Dongen JDM, Van Waes V, Venkatasubramanian G, Verdejo-Garcia A, Verveer I, Welsh JW, Wesley MJ, Witkiewitz K, Yavari F, Zarrindast MR, Zawertailo L, Zhang X, Cha YH, George TP, Frohlich F, Goudriaan AE, Fecteau S, Daughters SB, Stein EA, Fregni F, Nitsche MA, Zangen A, Bikson M, Hanlon CA. Transcranial electrical and magnetic stimulation (tES and TMS) for addiction medicine: A consensus paper on the present state of the science and the road ahead. Neurosci Biobehav Rev. 2019 Sep;104:118-140. doi: 10.1016/j.neubiorev.2019.06.007. Epub 2019 Jul 2. PMID 31271802
- [Background] Miron JP, Jodoin VD, Lesperance P, Blumberger DM. Repetitive transcranial magnetic stimulation for major depressive disorder: basic principles and future directions. Ther Adv Psychopharmacol. 2021 Sep 23;11:20451253211042696. doi: 10.1177/20451253211042696. eCollection 2021. PMID 34589203
- [Background] Zhang JJQ, Fong KNK, Ouyang RG, Siu AMH, Kranz GS. Effects of repetitive transcranial magnetic stimulation (rTMS) on craving and substance consumption in patients with substance dependence: a systematic review and meta-analysis. Addiction. 2019 Dec;114(12):2137-2149. doi: 10.1111/add.14753. Epub 2019 Aug 16. PMID 31328353
- [Background] Seewoo BJ, Hennessy LA, Jaeschke LA, Mackie LA, Etherington SJ, Dunlop SA, Croarkin PE, Rodger J. A Preclinical Study of Standard Versus Accelerated Transcranial Magnetic Stimulation for Depression in Adolescents. J Child Adolesc Psychopharmacol. 2022 Apr;32(3):187-193. doi: 10.1089/cap.2021.0100. Epub 2021 Dec 31. PMID 34978846
- [Background] Pushparaj A, Hamani C, Yu W, Shin DS, Kang B, Nobrega JN, Le Foll B. Electrical stimulation of the insular region attenuates nicotine-taking and nicotine-seeking behaviors. Neuropsychopharmacology. 2013 Mar;38(4):690-8. doi: 10.1038/npp.2012.235. Epub 2012 Nov 15. PMID 23249816
- [Background] Moretti J, Poh EZ, Rodger J. rTMS-Induced Changes in Glutamatergic and Dopaminergic Systems: Relevance to Cocaine and Methamphetamine Use Disorders. Front Neurosci. 2020 Mar 6;14:137. doi: 10.3389/fnins.2020.00137. eCollection 2020. PMID 32210744
- [Background] Lefaucheur JP, Aleman A, Baeken C, Benninger DH, Brunelin J, Di Lazzaro V, Filipovic SR, Grefkes C, Hasan A, Hummel FC, Jaaskelainen SK, Langguth B, Leocani L, Londero A, Nardone R, Nguyen JP, Nyffeler T, Oliveira-Maia AJ, Oliviero A, Padberg F, Palm U, Paulus W, Poulet E, Quartarone A, Rachid F, Rektorova I, Rossi S, Sahlsten H, Schecklmann M, Szekely D, Ziemann U. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS): An update (2014-2018). Clin Neurophysiol. 2020 Feb;131(2):474-528. doi: 10.1016/j.clinph.2019.11.002. Epub 2020 Jan 1. PMID 31901449
- [Background] Malik S, Jacobs M, Cho SS, Boileau I, Blumberger D, Heilig M, Wilson A, Daskalakis ZJ, Strafella AP, Zangen A, Le Foll B. Deep TMS of the insula using the H-coil modulates dopamine release: a crossover [11C] PHNO-PET pilot trial in healthy humans. Brain Imaging Behav. 2018 Oct;12(5):1306-1317. doi: 10.1007/s11682-017-9800-1. PMID 29170944
- [Background] McGirr A, Karmani S, Arsappa R, Berlim MT, Thirthalli J, Muralidharan K, Yatham LN. Clinical efficacy and safety of repetitive transcranial magnetic stimulation in acute bipolar depression. World Psychiatry. 2016 Feb;15(1):85-6. doi: 10.1002/wps.20300. No abstract available. PMID 26833619
- [Background] Dobek CE, Blumberger DM, Downar J, Daskalakis ZJ, Vila-Rodriguez F. Risk of seizures in transcranial magnetic stimulation: a clinical review to inform consent process focused on bupropion. Neuropsychiatr Dis Treat. 2015 Nov 30;11:2975-87. doi: 10.2147/NDT.S91126. eCollection 2015. PMID 26664122
- [Background] Keel JC, Smith MJ, Wassermann EM. A safety screening questionnaire for transcranial magnetic stimulation. Clin Neurophysiol. 2001 Apr;112(4):720. doi: 10.1016/s1388-2457(00)00518-6. No abstract available. PMID 11332408
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] McClintock SM, Reti IM, Carpenter LL, McDonald WM, Dubin M, Taylor SF, Cook IA, O'Reardon J, Husain MM, Wall C, Krystal AD, Sampson SM, Morales O, Nelson BG, Latoussakis V, George MS, Lisanby SH; National Network of Depression Centers rTMS Task Group; American Psychiatric Association Council on Research Task Force on Novel Biomarkers and Treatments. Consensus Recommendations for the Clinical Application of Repetitive Transcranial Magnetic Stimulation (rTMS) in the Treatment of Depression. J Clin Psychiatry. 2018 Jan/Feb;79(1):16cs10905. doi: 10.4088/JCP.16cs10905. PMID 28541649